CLINICAL TRIAL: NCT05613387
Title: A Randomized, Multiple Ascending Dose Trial Assessing Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of ZP8396 Administered to Healthy Subjects
Brief Title: A Research Study Looking at the Safety of Multiple Doses of ZP8396 and How it Works in the Body of Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zealand Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZP8396-21038
Record Dates: First submitted 2022-10-28; First posted 2022-11-14 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Overweight; Healthy Volunteers; Obese
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: Part 1: A single-centre, placebo-controlled, double-blind (within cohorts), randomised multiple ascending dose trial.
  Part 2: A single-centre, placebo-controlled, double-blind (within cohorts), randomised multiple ascending dose trial, using dose up-titration.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ZP8396 (Experimental): Part 1: 2 dose cohorts are planned with 10 subjects in each; 7 participants in each cohort will receive active treatment.
  Part 2: 3 dose cohorts are planned with 16 subjects in each; 12 participants in each cohort will receive active treatment.
  Interventions: Drug: ZP8396
- Placebo (ZP8396) (Placebo Comparator): Part 1: In each of the 2 dose cohorts, 3 subjects will receive placebo.
  Part 2: In each of the 3 cohorts, 4 subjects will receive placebo.
  Interventions: Drug: Drug: Placebo (ZP8396)

INTERVENTIONS:
Drug: ZP8396 — Part 1: Participants will receive 6 once-weekly doses of ZP8396 given subcutaneously (s.c., under the skin). Dose level will depend on the cohort.
  Part 2: Participants will receive 16 once-weekly doses of ZP8396 given subcutaneously (s.c., under the skin). Dose level will depend on the cohort. Dose up-titration will be used.
  Arms: ZP8396
Drug: Drug: Placebo (ZP8396) — Part 1: Participants will receive 6 once-weekly doses of placebo given subcutaneously (s.c., under the skin).
  Part 2: Participants will receive 16 once-weekly doses of placebo given subcutaneously (s.c., under the skin).
  Arms: Placebo (ZP8396)

SUMMARY:
The trial is a single-centre, randomised and double-blind within cohorts, placebo-controlled, sequential multiple ascending dose trial in normal weight and overweight but otherwise healthy subjects randomised to subcutaneous administration of ZP8396 or placebo

DETAILED DESCRIPTION:
The research study will investigate the safety and tolerability of ZP8396 in healthy study participants. In addition, the study will investigate how ZP8396 works in the body (pharmacokinetics and pharmacodynamics).

The trial is divided in two parts:

Part 1: 20 Participants will receive 6 once-weekly doses as an injection under the skin (subcutaneous, s.c.). Participants will have 14 visits with the study team. 6 of these visits consists of overnight stays of different duration (2-4 nights) at the study site. For each participant, the study will last up to 116 days.

Part 2: 48 Participants will receive 16 once-weekly doses as an injection under the skin (subcutaneous, s.c.) in a dose up-titration dose scheme. Participants will have 23 or 24 visits with the study team. 13 of these visits consists of overnight stays of different duration (2-4 nights) at the study site. For each participant, the study will last up to 198 days.

ELIGIBILITY:
Inclusion Criteria:

Part 1:

* Body Mass Index (BMI) between 21.0 and 29.9 kg/m^2, both inclusive
* Glycosylated hemoglobin (HbA1c) below 5.7 percent

Further inclusion criteria apply

Part 2:

* Body Mass Index (BMI) between 27.0 and 39.9 kg/m^2, both inclusive
* Glycosylated hemoglobin (HbA1c) below 6.5 percent

Further inclusion criteria apply

Exclusion Criteria:

Part 1:

* History of metabolic diseases more frequently associated with obesity, e.g. type-2-diabetes mellitus, hypertension, dyslipidemia, heart disease or stroke
* Systolic blood pressure below 90 mmHg or above 139 mmHg and/or diastolic blood pressure below 50 mmHg or above 89 mmHg
* Symptoms of arterial hypotension

Further exclusion criteria apply

Part 2:

* History of metabolic diseases more frequently associated with obesity, e.g. type-2-diabetes mellitus, hypertension, dyslipidemia, heart disease or stroke
* Systolic blood pressure below 90 mmHg or above 159 mmHg and/or diastolic blood pressure below 50 mmHg or above 99 mmHg
* Symptoms of arterial hypotension

Further exclusion criteria apply

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2022-11-07 (Actual); Primary Completion 2024-06-13 (Actual); Study Completion 2024-06-13 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events (TEAEs) | Part 1: From dosing (Day 1) to end of trial (Day 92); Part 2: From dosing (Day 1) to end of trial (Day 169 for Cohort 1 and 2, Day 176 for Cohort 3)
  Incidence of TEAEs from 1st dosing day to end of trial

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of ZP8396 (AUCτ) | Part 1: Day 1 (pre-dose) to Day 92; Part 2: Day 1 (pre-dose) to Day 169 for Cohort 1 and 2, Day 176 for Cohort 3
  Area under the plasma concentration-time curve over a dosing interval. Samples will be taken at set time points throughout the trial.
Pharmacokinetics (PK) of ZP8396 (AUCinf) | Part 1: Day 1 (pre-dose) to Day 92; Part 2: Day 1 (pre-dose) to Day 169 for Cohort 1 and 2, Day 176 for Cohort 3
  Area under the plasma concentration-time curve from time zero to infinity. Samples will be taken at set time points throughout the trial.
Pharmacokinetics (PK) of ZP8396 (AUClast) | Part 1: Day 1 (pre-dose) to Day 92; Part 2: Day 1 (pre-dose) to Day 169 for Cohort 1 and 2, Day 176 for Cohort 3
  Area under the plasma concentration-time curve from time zero to the time of the last measurable concentration. Samples will be taken at set time points throughout the trial.
Pharmacokinetics (PK) of ZP8396 (Cmax) | Part 1: Day 1 (pre-dose) to Day 92; Part 2: Day 1 (pre-dose) to Day 169 for Cohort 1 and 2, Day 176 for Cohort 3
  Maximum (peak) plasma drug concentration
Pharmacokinetics (PK) of ZP8396 (tmax) | Part 1: Day 1 (pre-dose) to Day 92; Part 2: Day 1 (pre-dose) to Day 169 for Cohort 1 and 2, Day 176 for Cohort 3
  Time to reach maximum (peak) plasma concentration
Pharmacokinetics (PK) of ZP8396 (λz) | Part 1: Day 1 (pre-dose) to Day 92; Part 2: Day 1 (pre-dose) to Day 169 for Cohort 1 and 2, Day 176 for Cohort 3
  Elimination rate constant
Pharmacokinetics (PK) of ZP8396 (t½) | Part 1: Day 1 (pre-dose) to Day 92; Part 2: Day 1 (pre-dose) to Day 169 for Cohort 1 and 2, Day 176 for Cohort 3
  Elimination half-life
Pharmacokinetics (PK) of ZP8396 (Vz/f) | Part 1: Day 1 (pre-dose) to Day 92; Part 2: Day 1 (pre-dose) to Day 169 for Cohort 1 and 2, Day 176 for Cohort 3
  Apparent volume of distribution
Pharmacokinetics (PK) of ZP8396 (CL/f) | Part 1: Day 1 (pre-dose) to Day 92; Part 2: Day 1 (pre-dose) to Day 169 for Cohort 1 and 2, Day 176 for Cohort 3
  Apparent total clearance of the drug from plasma
Pharmacokinetics (PK) of ZP8396 (Ctrough) | Part 1: Day 1 (pre-dose) to Day 92; Part 2: Day 1 (pre-dose) to Day 169 for Cohort 1 and 2, Day 176 for Cohort 3
  Trough concentration measured pre-dose
Accumulation Ratio for AUCτ | Part 1: Day 1 (pre-dose) to Day 92
  Accumulation Ratio for AUCτ
Accumulation Ratio for Cmax | Part 1: Day 1 (pre-dose) to Day 92
  Accumulation Ratio for Cmax
Pharmacodynamics (PD) of ZP8396 (Cmax acetaminophen) | Part 1: 0-240 minutes, relative to ingestion of MTM/acetaminophen on Day -1 (baseline), Day 5 and Day 40; Part 2: 0-240 minutes, relative to ingestion of MTM/acetaminophen on Day -1, Day 110 for cohort 1 and 2, Day -1, Day 1, Day 107 for cohort 3
  Maximum acetaminophen concentration after ingestion of a standardised Mixed Test Meal (MTM) and 1000 mg acetaminophen
Pharmacodynamics (PD) of ZP8396 (Tmax acetaminophen) | Part 1: 0-240 minutes, relative to ingestion of MTM/acetaminophen on Day -1 (baseline), Day 5 and Day 40; Part 2: 0-240 minutes, relative to ingestion of MTM/acetaminophen on Day -1, Day 110 for cohort 1 and 2, Day -1, Day 1, Day 107 for cohort 3
  Time to maximum acetaminophen concentration after ingestion of a standardised Mixed Test Meal (MTM) and 1000 mg acetaminophen
Pharmacodynamics (PD) of ZP8396 (AUCacetaminophen, 0-60 min) | Part 1: 0-60 minutes, relative to ingestion of MTM/acetaminophen on Day -1 (baseline), Day 5 and Day 40; Part 2: 0-60 minutes, relative to ingestion of MTM/acetaminophen on Day -1, Day 110 for cohort 1 and 2, Day -1, Day 1, Day 107 for cohort 3
  Area under the acetaminophen concentration-time curve from 0 to 60 minutes after ingestion of a standardised Mixed Test Meal (MTM) and 1000 mg acetaminophen
Pharmacodynamics (PD) of ZP8396 (AUCacetaminophen, 0-240 min) | Part 1: 0-240 minutes, relative to ingestion of MTM/acetaminophen on Day -1 (baseline), Day 5 and Day 40; Part 2: 0-240 minutes, relative to ingestion of MTM/acetaminophen on Day -1, Day 110 for cohort 1 and 2, Day -1, Day 1, Day 107 for cohort 3
  Area under the acetaminophen concentration-time curve from 0 to 240 minutes after ingestion of a standardised Mixed Test Meal (MTM) and 1000 mg acetaminophen
Pharmacodynamics (PD) of ZP8396 (Emax, Plasma Glucose [PG]) | Part 1: 0-240 minutes, relative to ingestion of MTM/acetaminophen on Day -1 (baseline), Day 5 and Day 40; Part 2: 0-240 minutes, relative to ingestion of MTM/acetaminophen on Day -1, Day 110 for cohort 1 and 2, Day -1, Day 1, Day 107 for cohort 3
  Maximum PG concentration from 0 to 240 minutes after ingestion of a standardised Mixed Test Meal (MTM) and 1000 mg acetaminophen
Pharmacodynamics (PD) of ZP8396 (Tmax, Plasma Glucose [PG]) | Part 1: 0-240 minutes, relative to ingestion of MTM/acetaminophen on Day -1 (baseline), Day 5 and Day 40; Part 2: 0-240 minutes, relative to ingestion of MTM/acetaminophen on Day -1, Day 110 for cohort 1 and 2, Day -1, Day 1, Day 107 for cohort 3
  Time to maximum PG concentration from 0 to 240 minutes after ingestion of a standardised Mixed Test Meal (MTM) and 1000 mg acetaminophen
Pharmacodynamics (PD) of ZP8396 (AUE, Plasma Glucose [PG], 0-60 minutes) | Part 1: 0-60 minutes, relative to ingestion of MTM/acetaminophen on Day -1 (baseline), Day 5 and Day 40; Part 2: 0-60 minutes, relative to ingestion of MTM/acetaminophen on Day -1, Day 110 for cohort 1 and 2, Day -1, Day 1, Day 107 for cohort 3
  Area under the acetaminophen concentration-time curve from 0 to 60 minutes after ingestion of a standardised Mixed Test Meal (MTM) and 1000 mg acetaminophen
Pharmacodynamics (PD) of ZP8396 (AUE, Plasma Glucose [PG], 0-240 minutes) | Part 1: 0-240 minutes, relative to ingestion of MTM/acetaminophen on Day -1 (baseline), Day 5 and Day 40; Part 2: 0-240 minutes, relative to ingestion of MTM/acetaminophen on Day -1, Day 110 for cohort 1 and 2, Day -1, Day 1, Day 107 for cohort 3
  Area under the acetaminophen concentration-time curve from 0 to 240 minutes after ingestion of a standardised Mixed Test Meal (MTM) and 1000 mg acetaminophen
Pharmacodynamics (PD) of ZP8396 (Emax, insulin) | Part 1: 0-240 minutes, relative to ingestion of MTM/acetaminophen on Day -1 (baseline), Day 5 and Day 40
  Maximum insulin concentration from 0 to 240 minutes after ingestion of a standardised Mixed Test Meal (MTM) and 1000 mg acetaminophen
Pharmacodynamics (PD) of ZP8396 (Tmax, insulin) | Part 1: 0-240 minutes, relative to ingestion of MTM/acetaminophen on Day -1 (baseline), Day 5 and Day 40
  Time to maximum insulin concentration from 0 to 240 minutes after ingestion of a standardised Mixed Test Meal (MTM) and 1000 mg acetaminophen
Pharmacodynamics (PD) of ZP8396 (AUEinsulin,0-60 minutes) | Part 1: 0-60 minutes, relative to ingestion of MTM/acetaminophen on Day -1 (baseline), Day 5 and Day 40
  Area under the insulin concentration-time curve from 0 to 60 minutes after ingestion of a standardised Mixed Test Meal (MTM) and 1000 mg acetaminophen
Pharmacodynamics (PD) of ZP8396 (AUEinsulin,0-240 min) | Part 1: 0-240 minutes, relative to ingestion of MTM/acetaminophen on Day -1 (baseline), Day 5 and Day 40
  Area under the insulin concentration-time curve from 0 to 240 minutes after ingestion of a standardised Mixed Test Meal (MTM) and 1000 mg acetaminophen
Pharmacodynamics (PD) of ZP8396 (Emax, glucagon) | Part 1: 0-240 minutes, relative to ingestion of MTM/acetaminophen on Day -1 (baseline), Day 5 and Day 40
  Maximum glucagon concentration from 0 to 240 minutes after ingestion of a standardised Mixed Test Meal (MTM) and 1000 mg acetaminophen
Pharmacodynamics (PD) of ZP8396 (Tmax, glucagon) | Part 1: 0-240 minutes, relative to ingestion of MTM/acetaminophen on Day -1 (baseline), Day 5 and Day 40
  Time to maximum glucagon concentration from 0 to 240 minutes after ingestion of a standardised Mixed Test Meal (MTM) and 1000 mg acetaminophen
Pharmacodynamics (PD) of ZP8396 (AUEglucagon,0-60 minutes) | Part 1: 0-60 minutes, relative to ingestion of MTM/acetaminophen on Day -1 (baseline), Day 5 and Day 40
  Area under the glucagon concentration-time curve from 0 to 60 minutes after ingestion of a standardised Mixed Test Meal (MTM) and 1000 mg acetaminophen
Pharmacodynamics (PD) of ZP8396 (AUEglucagon,0-240 minutes) | Part 1: 0-240 minutes, relative to ingestion of MTM/acetaminophen on Day -1 (baseline), Day 5 and Day 40
  Area under the glucagon concentration-time curve from 0 to 240 minutes after ingestion of a standardised Mixed Test Meal (MTM) and 1000 mg acetaminophen

CONTACTS AND LOCATIONS:
Overall Officials: Zealand Pharma A/S, Study Director — Zealand Pharma A/S
Locations (1):
- Profil Institut für Stoffwechselforschung GmbH, Neuss, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No